CLINICAL TRIAL: NCT05877092
Title: Comparative Evaluation of Masticatory Efficiency of Implant Supported Thermoplastic Versus Conventional Acrylic Resin Mandibular Overdenture With Bar/Clip Attachment
Brief Title: Comparative Evaluation of Masticatory Efficiency of Implant Supported Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hamada Zaki Mahross Atia, Assistant Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 903/2935
Record Dates: First submitted 2023-05-06; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Mastication Disorder; Mandibular Dysfunction
Keywords: Masticatory efficiency; thermoplastic base material; Bar attachment system
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Denture, Overlay

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acrylic resin denture base (Active Comparator): complete overdenture constructed from heat cured acrylic resin for Group I
  Interventions: Device: implants with overdentures
- thermoplastic denture (Active Comparator): complete thermoplastic denture was constructed for Group II
  Interventions: Device: implants with overdentures

INTERVENTIONS:
Device: implants with overdentures — two implants with bar attachment placed in interforaminal of the mandible mandible of the participants, the patients were delivered conventional upper complete denture constructed from heat cured acrylic rein, but in implanted mandibular arch they were received complete overdenture constructed from heat cured acrylic resin for Group I, and complete thermoplastic denture was constructed for Group II.

SUMMARY:
the goal of this clinical trial To evaluate the effects of different base materials of mandibular implant supported overdenture with bar/clip attachment on masticatory efficacy.

Twenty-four edentulous patients were selected to place two inter-foraminal mandibular implants with custom-made cast bar to retain overdentures made from two different base material and divided into two groups.

The masticatory efficiency were tested using three different food categories (carrots, bananas, and apples) and measured by four parameters.

DETAILED DESCRIPTION:
Based on inclusion and exclusion standards for implant selection, a twenty-four completely edentulous medically fit male patient aged 50-70 years were selected from the removable prosthodontics clinical, Faculty of Dental Medicine. The patient selection was determined through oral and dental examination, which revealed class I arch relationship with adequate 20-25MM inter-arch space and free from any oral hard or soft tissue abnormality that can interfere with the treatment. The selection was excluded all patients who do not satisfy these normal criteria. Written consent was obtained from each patients, detailing all surgical and prosthetic steps as well as the treatment's advantages and disadvantages.

To obtain precise measurements of bone height and width at the implant site and accurately determine the size and type of the required implants, Cone Beam Computerized Tomography (CBCT) was performed, guided with a radiographic stent for each selected patient.

According to the type of complete denture base material's construction, the twenty-four selected patients whose selected to participate in this trial, were grouped into two groups. Group I (n =12) patients with a heat polymerized acrylic resin complete mandibular overdenture HCG and In Group II (n =12) patients with a thermoplastic (polyamide) complete mandibular overdenture TPG, both groups were retained by a bar/clip attachment system.

The masticatory efficiencies were examined using three different food categories in terms of the level of hardness, such as (apples, bananas, and carrots). Patients installed their mandibular overdentures while sitting upright. Each participant was then given assurances to help them rest and not be disturbed before eating the test food, which was cut into equal parts (1cm × 1cm). The following measures were recorded using a stopwatch:

The Number of chewing cycle strokes up to the first sallow. The Number of chewing cycle strokes until the mouth is free of food. The number of swallows until the mouth is free of food. Time (in seconds) until the mouth is free of food. The data collected from the test groups, and a statistical evaluation conducted using the SPSS software program (IBM Company). The average, standard deviation, and lowest and highest values were also calculated for each group under consideration. A one-way ANOVA was also used to ascertain whether there were any significant differences in the averages of the different groups analyzed. Additionally, the Tukey test was used to evaluate whether averages differed significantly from each other at the specific probability level (P < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous
* class I arch relationship
* 20-25MM inter-arch space
* free from any oral hard or soft tissue abnormality

Exclusion Criteria:

* partially dentate patients
* abnormal arch class (class II or III)
* patients wit flabby tissue, acquired defects, or bony exccestosis.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Completely edentulous medically fit male patient aged 50-70 years
Enrollment: 24 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Test of Masticatory Efficiency by using three different food categories | immediately after dentures were placed.
  The masticatory efficiencies were examined using three different food categories in terms of the level of hardness, such as (apples, bananas, and carrots).
The Number of chewing cycle strokes up to the first sallow | immediately after dentures placed.
  by using a stopwatch, The Number of chewing cycle strokes up to the first sallow recorded
The Number of chewing cycle strokes until the mouth is free of food | immediately after dentures placed.
  by using a stopwatch, The Number of chewing cycle strokes until the mouth is free of food recorded
The number of swallows until the mouth is free of food | immediately after dentures placed.
  by using a stopwatch, The number of swallows until the mouth is free of food
Time (in seconds) until the mouth is free of food | immediately after dentures placed.
  by using a stopwatch, Time (in seconds) until the mouth is free of food

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No